CLINICAL TRIAL: NCT04656522
Title: A Participatory Comic Intervention for Sexual Violence Prevention and Post-rape Care With Refugee Adolescents and Youth in a Humanitarian Setting in Uganda
Brief Title: Comic Intervention for Sexual Violence Prevention and Post-rape Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Carmen Logie, MSW, PhD, Associate Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: gcc_bidibidi
Record Dates: First submitted 2020-11-13; First posted 2020-12-07 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Knowledge, Attitudes, Practice; Post-exposure Prophylaxis
Keywords: Digital health intervention; Forcibly displaced youth; Uganda; Post-exposure prophylaxis; Bystander practices; Sexual Violence Stigma; Gender based violence
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: A single-arm, pre-test/post-test trial design will be used to evaluate the effectiveness of a participatory comic intervention on changes in PEP knowledge and acceptability, sexual violence stigma, and bystander beahviour with displaced/refugee youth and health care providers in Bidi Bidi Refugee Settlement, Uganda.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participatory Comic Intervention (Experimental): This is a pre-test/post-test trial, therefore all participants will participate in the participatory comic intervention.
  Interventions: Behavioral: Participatory Comic Intervention

INTERVENTIONS:
Behavioral: Participatory Comic Intervention — This participatory comic intervention promotes sexual violence prevention and post-rape care with refugee youth and health care providers. In 4-hour workshops, a customized comic book featuring eight sexual violence scenarios will be distributed. Each 1-page scenario speaks to a unique theme of sexual violence experiences among youth or post-rape care preferences. During the workshop participants will explore social, sexual, and psychological needs of youth in Bidi Bidi and practice ways of developing and maintaining healthy relationships (youth) as well as discuss post-rape care responses that attend to the needs and priorities of young refugees in Bidi Bidi who have experienced sexual violence (health care providers). Each workshop will include 20 participants and will be facilitated by trained staff from Real Medicine, Uganda. Further, each workshop will have at least 2 facilitators who are trained in the bystander model.

SUMMARY:
In humanitarian settings, sexual and gender-based violence disproportionately impacts women and children. However, there continues to be a lack of evidence regarding both sexual violence prevention and post-rape care interventions in low- and middle-income humanitarian contexts, with even less evidence supporting adolescents and youth in these settings. Participatory comics offer a youth-friendly, low-cost, scalable approach for preventing sexual violence and training clinicians in post-rape care in humanitarian settings. This study aims to develop, implement, and evaluate the effectiveness of a comic intervention on preventing sexual violence and improving post-rape care with youth aged 16-24 and health care providers in the Bidi Bidi refugee settlement.

DETAILED DESCRIPTION:
Uganda is Sub-Saharan Africa's largest refugee host community; with over 250,000 residents, Bidi Bidi is the largest refugee settlement in Uganda and the second largest globally. In humanitarian settings, sexual and gender-based violence disproportionately impacts women and children. However, there continues to be a lack of evidence regarding both sexual violence prevention and post-rape care interventions in low- and middle-income humanitarian contexts, with even less evidence supporting adolescents and youth in these settings. Stigma directed toward adolescent sexual practices and engagement in sexual and reproductive health services, such as contraception, HIV testing, and post-exposure prophylaxis (PEP), is also associated with social isolation, violence and mental health challenges. Participatory comics offer a youth-friendly, low-cost, scalable approach for preventing sexual violence and training clinicians in post-rape care in humanitarian settings. This study aims to develop, implement, and evaluate the effectiveness of a comic intervention on preventing sexual violence and improving post-rape care with youth aged 16-24 and health care providers in the Bidi Bidi refugee settlement. Participating youth and health care providers will take part in 4-hour peer-facilitated workshops exploring topics of social, sexual, and psychological needs and pro-social interventions (youth) and post-rape care responses and attending to the needs of youth refugees who have experienced sexual violence (health care providers) using comics developed with qualitative data collected from an earlier study phase. Using a pre-test/post-test design, this study will assess changes in participants' PEP knowledge and acceptance, bystander behaviour, and sexual violence stigma.

ELIGIBILITY:
Inclusion Criteria (Youth):

* Resides in Bidi Bidi Refugee Settlement Zone 3
* Identify as a refugee/displaced person
* Aged 16-24 years
* Speak English, Bari or Arabic

Exclusion Criteria (Youth):

* Does not reside in Bidi Bidi Refugee Settlement Zone 3
* Does not identify as a refugee/displaced person
* Is less than age 16 years or older than age 24 years
* Does not speak English, Bari or Arabic

Inclusion Criteria (Healthcare Provider):

* Provides healthcare services in Bidi Bidi Refugee Settlement and/or Yumbe, Uganda
* Aged greater than or equal to 18 years
* Speak English, Bari or Arabic

Exclusion Criteria (Healthcare Provider):

* Does not provide healthcare services in Bidi Bidi Refugee Settlement and/or Yumbe, Uganda
* Less than age 18 years
* Does not speak English, Bari or Arabic

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in PEP Knowledge & Acceptability | Time 1 (0-baseline), Time 2 ( 6 hours follow-up), Time 3 (4 week follow-up)
  PEP knowledge and acceptability assessed through testing participants on their knowledge of correct PEP use and asked to report on their acceptance towards PEP use and adherence. Scores are binary yes/no.
Changes in Bystander Practices | Time 1 (0-baseline), Time 2 ( 6 hours follow-up), Time 3 (4 week follow-up)
  Bystander practices assessed through the Bystander Decision Balance Scale and Slaby Bystander Efficacy Scale (Range 16-64). Higher scores indicate increased bystander practices.
Changes in Sexual Violence Stigma | Time 1 (0), Time 2 (5hours), Time 3 (4 weeks post-workshop)
  Attitudes and beliefs towards sexual violence will be assessed using the Sexual Violence Stigma scale (Range 17-68). Higher score indicates poorer attitudes and beliefs, and thus greater stigma, towards sexual violence and sexual violence survivors.

SECONDARY OUTCOMES:
Changes in Gender Equitable Norms | Time 1 (0-baseline), Time 2 ( 6 hours follow-up), Time 3 (4 week follow-up)
  Gender Equitable Norms will be assessed using the physical violence subscale (Range 6-18) of the gender equitable men (GEM) scale to measure attitudes towards gender equitable norms considering the prevailing norms in the community concerning physical violence. A higher score indicates positive attitudes towards gender equitable norms.
Changes in Depression | Time 1 (0-baseline), Time 3 (4 week follow-up)
  Depression outcomes will be assessed using the Patient Health Questionnaire 2-item (PHQ-2) (Range 0-6). Scores of 3 or above signal major depressive disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen H Logie, PhD, Principal Investigator — University of Toronto, Canada
Locations (2):
- Factor-Inwentash Faculty of Social Work, University of Toronto, Toronto, Ontario, Canada
- Uganda Refugee and Disaster Management Council, Arua, Uganda

REFERENCES:
- [Derived] Logie CH, Okumu M, Loutet M, Berry I, Lukone SO, Kisubi N, Mwima S, Kyambadde P. Mixed-methods findings from the Ngutulu Kagwero (agents of change) participatory comic pilot study on post-rape clinical care and sexual violence prevention with refugee youth in a humanitarian setting in Uganda. Glob Public Health. 2023 Jan;18(1):2092178. doi: 10.1080/17441692.2022.2092178. Epub 2022 Jun 30. PMID 35770702